CLINICAL TRIAL: NCT01869556
Title: Comparison of Intravenous Ergonovine With Intramuscular Carboprost, Both in Combination With Oxytocin Infusion, During Cesarean Section for Failure to Progress in Labor: A Double-blinded Placebo-controlled Randomized Controlled Trial
Brief Title: Comparison of IV Ergonovine With IM Carboprost, With Oxytocin IV, During Cesarean Section for Failure to Progress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-05
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; Cesarean delivery; failure to progress in labor
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Ergonovine; Carboprost; carboprost tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxytocin only (Active Comparator): Oxytocin 5IU IV bolus, followed by an infusion of oxytocin 20IU/L, running at at rate of 40mIU/min for 8 hours
  Interventions: Drug: Oxytocin
- Oxytocin + Ergot (Active Comparator): Oxytocin 5IU IV bolus + Ergot 0.25mg IV, followed by an infusion of oxytocin 20IU/L, running at at rate of 40mIU/min for 8 hours
  Interventions: Drug: Oxytocin; Drug: Ergot
- Oxytocin + Carboprost (Active Comparator): Oxytocin 5IU IV bolus + Carboprost 0.25mg IM, followed by an infusion of oxytocin 20IU/L, running at at rate of 40mIU/min for 8 hours
  Interventions: Drug: Oxytocin; Drug: Carboprost

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 5IU IV bolus, followed by an infusion of oxytocin 20IU/L, running at at rate of 40mIU/min for 8 hours
  Other Names: syntocinon
Drug: Ergot — Ergot 0.25mg IV
  Other Names: ergonovine maleate
  Arms: Oxytocin + Ergot
Drug: Carboprost — Carboprost 0.25mg IM
  Other Names: Hemabate®
  Arms: Oxytocin + Carboprost

SUMMARY:
Patients having Cesarean section after they have been in labor for many hours bleed much more, in average twice as much, as compared with patients having an elective Cesarean section. The investigators believe a simple change in practice might contribute to reduce this bleeding. This study will involve the use of oxytocin (also known as syntocinon), ergonovine (also known as ergot) and carboprost (also known as hemabate). Oxytocin is routinely used to help contract the uterus and keep it contracted after the delivery of the baby and placenta, so as to reduce the amount of blood loss. Ergonovine is also given through the intravenous line, while carboprost is given as an injection in the muscle. Although they are not routinely given in every case, these are very frequently given as rescue medications to patients who fail to respond appropriately to oxytocin. This study is designed to determine if ergonovine or carboprost given in association with oxytocin, in a preventive way, after delivery of the baby and placenta, can reduce the amount of blood loss during Cesarean sections following a trial of labour.

DETAILED DESCRIPTION:
The objective of the investigators study is to compare the efficacy of intravenous ergonovine and intramuscular carboprost, when administered with oxytocin infusion, prophylactically to decrease blood loss at Cesarean section for labor arrest. Desensitization of the oxytocin receptors has been recently demonstrated in cultured human myometrial cells after continuous and prolonged exposure to oxytocin in-vitro. This could be also the reason for a greater risk of uterine atony and postpartum hemorrhage (PPH) seen in women requiring induction and augmentation of labor. Therefore, addition of a different uterotonic agent, involving a different mechanism of action, to oxytocin infusion is likely to be beneficial, especially in women undergoing CS following failure to progress in labor, who are at a greater risk for PPH.

ELIGIBILITY:
Inclusion Criteria:

* patients who give written informed consent
* patients undergoing Cesarean section for failure to progress in labour, under regional anesthesia
* patients should be in the first stage of labour and have received oxytocin for at least 4 hours

Exclusion Criteria:

* patients who refuse to give written informed consent
* patients who require general anesthesia
* patients who claim allergy or hypersensitivity to oxytocin, ergot derivatives or prostaglandins
* patients with cardiac diseases and hypertension or preeclampsia ( diastolic blood pressure > 90 mmHg, systolic blood pressure > 140 mmHg )
* patients with asthma or any other respiratory disease
* patients with conditions at risk of PPH such as placenta previa, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, previous history of uterine atony and postpartum bleeding, bleeding diathesis and known infection.

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2013-06-04 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Need for additional uterotonics intraoperatively | 1 hour
  Need for additional uterotonics intraoperatively if requested by the surgeon, YES or NO

SECONDARY OUTCOMES:
Effectiveness of uterine contraction | 10 min
  Adequate/inadequate uterine tone at 3,5 & 10 min
Need for blood transfusion | 24 hours
  Any blood products administered
Vital signs | 2 hours
  In the OR, heart rate, blood pressure, and oxygen saturation will be measured and looked at for abnormalities
Side effects | 24 hours
  The presence of nausea, vomiting,other dysrhythmias, chest pain, headache, bronchospasm and any others will be recorded.
Estimated blood loss | 48 hours
  calculated blood loss = EBV (Pre-op Htc-Post-op Htc) EBV (estimated blood volume, mL)=patient's weight in kg x 85
Need for additional uterotonics or interventions post-operatively | 24 hours
  Need for additional uterotonics or interventions post-operatively up to 24 hours post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Balki M, Downey K, Walker A, Seaward G, Carvalho JCA. Prophylactic Administration of Uterotonics to Prevent Postpartum Hemorrhage in Women Undergoing Cesarean Delivery for Arrest of Labor: A Randomized Controlled Trial. Obstet Gynecol. 2021 Mar 1;137(3):505-513. doi: 10.1097/AOG.0000000000004288. PMID 33543897